CLINICAL TRIAL: NCT01716455
Title: A Phase 1, Open-label, Single-dose Study of the Pharmacokinetics, Safety, and Tolerability of SSP-004184 (FBS0701) in Healthy Adults and Elderly Subjects and in Subjects With Impaired Renal Function
Brief Title: Study of SSP-004184 (FBS0701) in Healthy Adults and Elderly Subjects and in Subjects With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPD602-104
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Results first posted 2014-02-19 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Impaired Renal Function
MeSH Terms: conditions — Renal Insufficiency | interventions — 4,5-dihydro-2-(2-hydroxy-3-(3,6,9-trioxadecyloxy)phenyl)-4-methyl-4-thiazolecarboxylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- SSP-004184 (Mild Renal Impairment) (Experimental): All subjects will take a single dose of SSP-004184 (75 mg/kg, oral capsule) on Day 1
  Interventions: Drug: SSP-004184
- SSP-004184 (Moderate Renal Impairment) (Experimental): All subjects will take a single dose of SSP-004184 (75 mg/kg, oral capsule) on Day 1
  Interventions: Drug: SSP-004184
- SSP-004184 (Severe Renal Impairment) (Experimental): All subjects will take a single dose of SSP-004184 (75 mg/kg, oral capsule) on Day 1
  Interventions: Drug: SSP-004184
- SSP-004184 (End Stage Renal Disease) (Experimental): All subjects will take a single dose of SSP-004184 (75 mg/kg, oral capsule) on Day 1
  Interventions: Drug: SSP-004184
- SSP-004184 (Healthy Elderly Subjects) (Experimental): All subjects will take a single dose of SSP-004184 (75 mg/kg, oral capsule) on Day 1
  Interventions: Drug: SSP-004184
- SSP-004184 (Matched Healthy Subjects) (Experimental): All subjects will take a single dose of SSP-004184 (75 mg/kg, oral capsule) on Day 1. Healthy subjects matched to renally impaired subjects in arms 1 through 4. (Note: One healthy subject can match more than one renally impaired subject.)
  Interventions: Drug: SSP-004184

INTERVENTIONS:
Drug: SSP-004184
  Other Names: SPD602, FBS0701

SUMMARY:
Shire is developing SSP-004184 (FBS0701), a novel iron chelator , for the treatment of chronic iron overload in patients with transfusion-dependent hereditary and acquired anemias. The primary purpose of the study is to assess the pharmacokinetics of SSP-004184 (FBS0701) following a single 75mg/kg dose of SSP-004184 (FBS0701) in healthy adults and elderly subjects and in adult subjects with mild, moderate, severe, and end stage renal disease (ESRD) degrees of impaired renal function. The results of this study will characterize the pharmacokinetics, safety, and tolerability of SSP-004184 (FBS0701) in adult subjects with various degrees of renal impairment, and these data will be compared to healthy adult and elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects

* Age 18-85 years inclusive at the time of consent. The elderly treatment group will be defined by an age over 65 years. It is required that at least 4 of the subjects in the elderly group will be over 75 years old.
* All subjects will be "healthy"
* Normal renal function (in 18-65 year-old subjects), defined as an estimated glomerular filtration rate (eGFR) from the Modification of Diet in Renal Disease (MDRD) Study of >90 mL/min/ 1.73 m2 at the Screening Visit.
* The stability of renal function will be confirmed by 2 determinations of serum creatinine separated by at least 7 days

Subjects with renal impairment

* Age 18-85 years inclusive at the time of consent.
* Estimated glomerular filtration rate from the MDRD Study is to be estimated at the Screening Visit and should be as described in FDA guidance.
* Subjects must have no clinically significant abnormalities (except for abnormalities explained by the renal impairment disorder).

All subjects

* Willingness to comply with any applicable contraceptive requirements of the protocol and is:
* Male, or
* Non pregnant, non lactating female
* Females must be at least 90 days post partum or nulliparous.
* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6 (1996) and applicable regulations, before completing any study related procedures. The date of signing informed consent is defined as the beginning of the Screening Period
* Body mass index between 18.5-40.0 kg/m² inclusive. This inclusion criterion will only be assessed at the Screening Visit.
* Hemoglobin of 9.0 g/dL or greater at the Screening Visit and Day -2.
* No clinically significant deviations from the reference ranges for clinical laboratory tests as evaluated by the investigator. Low-density lipoprotein cholesterol value must be <189 mg/dL and triglycerides value must be <499 mg/dL at the Screening Visit.
* Ability to swallow a dose of investigational product.

Exclusion Criteria:

Healthy subjects

* Subject has a clinically significant history or a disorder detected during the medical interview/physical examination
* Current or relevant previous history of serious, severe or unstable (acute or progressive) physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
* History of diabetes mellitus, nephrotic syndrome (defined as plasma albumin <30 g/dL and/or proteinuria >3 g/day), or other metabolic endocrine disease known to be associated with alterations in plasma lipid levels. Uncontrolled hypothyroidism is defined as thyroid stimulating hormone (TSH) 1.5 times greater than the upper limit of normal (ULN).

Subjects with renal impairment

* Current or recurrent disease, other than impaired renal function that could affect, the action, absorption or disposition of the investigational product, or clinical or laboratory assessments.
* Concurrent chronic or acute illness or unstable medical condition (other than those associated with their renal disease) that may deteriorate and thus confound the results of safety assessments, increase risk to the subject or lead to difficulty complying with the protocol.
* A potassium concentration >6.2 mmol/L at the Screening Visit.
* Subjects with a renal transplant.
* History of nephrotic syndrome (defined as plasma albumin <30 g/dL and/or proteinuria >3 g/day), or other metabolic endocrine disease known to be associated with alterations in plasma lipid levels (uncontrolled hypothyroidism defined as TSH 1.5 times greater than the upper reference range value).
* Subjects on peritoneal dialysis.
* Uncontrolled systolic or diastolic blood pressure as defined by the investigator.
* Liver enzymes (ALT, AST, GGT) more than 2 fold above ULN at the Screening Visit or on Day -2.
* Uncontrolled diabetes mellitus as determined by the investigator.
* Congestive Heart Failure classified New York Heart Association (NYHA) Class III or IV.
* Any major illness that would in the opinion of the investigator put study subject at risk or interfere with study conduct.

All subjects

* Acute illness, as judged by the investigator, within 2 weeks of the first dose of investigational product.
* Known or suspected intolerance or hypersensitivity to the investigational products, closely related compounds, or any of the stated ingredients.
* Subject has a history of thyroid disorder that has not been stabilized on thyroid medication or treatment within 3 months of the Screening Visit.
* History of alcohol or other substance abuse within the last year.
* A positive screen for alcohol or drugs of abuse at the Screening Visit or on Day -2.
* Male subjects who consume more than 3 units of alcohol per day. Female subjects who consume more than 2 units of alcohol per day. One alcohol unit=1 beer (12 oz/355 mL) = 1 wine (5 oz/150 mL) = 1 liquor (1.5 oz/40 mL)
* A positive human immunodeficiency virus (HIV) antibody screen, Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibody screen.
* Current use of any other medication (including over-the-counter, herbal or homeopathic preparations) that could affect (improve or worsen) the condition being studied, or could affect the action, absorption, or disposition of the investigational product(s), or clinical or laboratory assessment. (Current use is defined as use within 14 days of dosing). Subjects must be on a stable dose of allowed medications for 14 days prior to dosing.
* Use of tobacco in any form (eg, smoking or chewing) or other nicotine-containing products in any form (eg, gum, patch) within 30 days prior to the first dose of investigational product.
* Routine consumption of more than 2 units of caffeine per day or subjects who experience caffeine withdrawal headaches or have a history of caffeine withdrawal headaches. (One caffeine unit is contained in the following items: one 6oz/180mL cup of coffee, two 12 oz/355 mL cans of cola, one 12 oz/355 mL cup of tea, three 1oz/28g chocolate bars. Decaffeinated coffee, tea, or cola are not considered to contain caffeine).
* Donation of blood or blood products (eg, plasma or platelets) within 60 days prior to the first dose of investigational product.
* Use of another investigational product within 30 days prior to receiving the first dose of investigational product or active enrollment in another drug or vaccine clinical study.
* Substantial changes in eating habits within 30 days prior to receiving the first dose of investigational product, as assessed by the investigator.
* An inability to follow a standardized diet and meal schedule or inability to fast, as required during the study.
* Prior screen failure, randomization, participation, or enrollment in this study.
* Any known hypersensitivity to iohexol or to iodine per se.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-10-29 (Actual); Primary Completion 2013-03-10 (Actual); Study Completion 2013-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center (OCRC), Orlando, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- SSP-004184 (Mild Renal Impairment); SSP-004184 (Moderate Renal Impairment); SSP-004184 (Severe Renal Impairment); SSP-004184 (End Stage Renal Disease); SSP-004184 (Matched Healthy Subjects); SSP-004184 (Healthy Elderly Subjects): All subjects took a single oral dose of SSP-004184 (75 mg/kg) on Day 1
Period: Overall Study
Arm/Group | SSP-004184 (Mild Renal Impairment) | SSP-004184 (Moderate Renal Impairment) | SSP-004184 (Severe Renal Impairment) | SSP-004184 (End Stage Renal Disease) | SSP-004184 (Matched Healthy Subjects) | SSP-004184 (Healthy Elderly Subjects)
Started | 8 | 8 | 8 | 8 | 26 | 8
Completed | 8 | 8 | 8 | 8 | 26 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SSP-004184 (Mild Renal Impairment) | SSP-004184 (Moderate Renal Impairment) | SSP-004184 (Severe Renal Impairment) | SSP-004184 (End Stage Renal Disease) | SSP-004184 (Matched Healthy Subjects) | SSP-004184 (Healthy Elderly Subjects) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 26 | 8 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (4.47) | 63.4 (7.56) | 64.4 (8.23) | 44.5 (5.58) | 55.6 (10.81) | 72.6 (5.29) | 58.7 (11.23)
Age, Customized [Count of Participants; unit: Participants]
  >=65 years | 0 | 3 | 5 | 0 | 6 | 8 | 22
  Between 18 and 65 years | 8 | 5 | 3 | 8 | 20 | 0 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 4 | 9 | 2 | 21
  Male | 6 | 6 | 6 | 4 | 17 | 6 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 8 | 8 | 8 | 8 | 26 | 8 | 66

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) of SSP-004184
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Over 96 hours post-dose
Population: The Pharmacokinetic Analysis Set is defined as all subjects in the Safety Analysis Set for whom the primary pharmacokinetic data are considered sufficient and interpretable. The Safety Analysis Set consists of all enrolled subjects who take at least 1 dose of investigational product and have at least 1 post dose safety assessment.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | SSP-004184 (Mild Renal Impairment) | SSP-004184 (Moderate Renal Impairment) | SSP-004184 (Severe Renal Impairment) | SSP-004184 (End Stage Renal Disease) | SSP-004184 (Matched Healthy Subjects) | SSP-004184 (Healthy Elderly Subjects)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 26 | 8
ng*hr/ml | 445892.7 (156768.3) | 932688.3 (413237.0) | 1531185.8 (836393.5) | 1261081.6 (611849.8) | 397400.1 (126991.1) | 559880.8 (208295.5)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of SSP-004184
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated.
Time Frame: Over 96 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SSP-004184 (Mild Renal Impairment) | SSP-004184 (Moderate Renal Impairment) | SSP-004184 (Severe Renal Impairment) | SSP-004184 (End Stage Renal Disease) | SSP-004184 (Matched Healthy Subjects) | SSP-004184 (Healthy Elderly Subjects)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 26 | 8
ng/ml | 157412.5 (39231.8) | 168362.5 (43300.5) | 158250.0 (34154.1) | 146562.5 (51181.4) | 136588.5 (40910.5) | 161525.0 (53088.4)

ADVERSE EVENTS:
Groups:
- Impaired Renal Function; Matched Healthy Subjects; Healthy Elderly Subjects: All subjects took a single oral dose of SSP-004184 (75 mg/kg) on Day 1
Arm/Group | Impaired Renal Function | Matched Healthy Subjects | Healthy Elderly Subjects
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/26 | 0/8
Other Adverse Events (participants affected / at risk) | 14/32 | 9/26 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Impaired Renal Function (N=32) | Matched Healthy Subjects (N=26) | Healthy Elderly Subjects (N=8)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Urine colour abnormal (Investigations) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Chromaturia (drug-induced urine coloration) (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Liver Function Test Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.